CLINICAL TRIAL: NCT03519529
Title: The Relationship Between Sex Hormone Binding Globulin, Testosterone and Glycemic Control in Patients With Type 2 Diabetes
Brief Title: Sex Hormone Binding Globulin, Testosterone and Glycemic Control in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: ENDO20180426-01
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Type2 Diabetes
Keywords: sex hormone-binding globulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sex hormone-binding globulin(SHBG) is a surrogate marker of insulin resistance. This study aims at the characteristic and clinical significance of SHBG and testosterone in patients with type 2 diabetes(T2D).

DETAILED DESCRIPTION:
The investigators recorded clinical factors, biochemical criterion such as serum levels of glucose and lipids, HbA1c, SHBG, testosterone, insulin, EPO, C-peptide, glucagon, microalbuminuria, glycemic variation via CGM, carotid plaque, ECG and ultrasonic cardiogram in patients with T2D who visited in the Department of Endocrinology at the Nanjing First Hospital from January 2015 to Aprol 2018. The relationship between levels of SHBG, testosterone and glycemic variation/diabetic complications are analysed.

ELIGIBILITY:
Inclusion Criteria:

● Patients with T2D and the diagnostic criteria of T2D is according to the World Health Organization in 1999.

Exclusion Criteria:

* Patients use systemic steroidal anti-inflammatory drugs.
* Patients with an acute infection.
* Patients with acute complication of diabetes.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes who visited in the Department of Endocrinology at the Nanjing First Hospital from January 2015 to April 2018 were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
sex hormone-binding globulin | Day 1
  the blood sex hormone-binding globulin level of patients

SECONDARY OUTCOMES:
Testosterone | Day 1
  blood testosterone level of patients
EPO | Day 1
  blood erythropoietin level of patients
HbA1c | Day 1
  the glycosylated hemoglobin level of patients
MBG | Day 1-4
  24h mean blood glucose tested by CGM
MAGE | Day 1-4
  the 24h mean amplitude of glycemic excursion
SD | Day 1-4
  the standard deviation of mean glucose

REFERENCES:
- [Derived] Ding B, Sun R, Zhai XF, Lu TT, Cheng L, Li FF, Hu Y, Ma JH. Association of high circulating testosterone with increased glycaemic variability in type 2 diabetes: A cross-sectional study in China. Diabetes Metab Res Rev. 2019 May;35(4):e3126. doi: 10.1002/dmrr.3126. Epub 2019 Jan 23. PMID 30614187